CLINICAL TRIAL: NCT03211806
Title: Technology to Reduce Sedentary Behavior Before and After Cancer Surgery
Brief Title: Detecting Activity to Support Healing
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carissa Low, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-075; K07CA204380 (NIH)
Record Dates: First submitted 2017-01-23; First posted 2017-07-07 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer; Peritoneal Cancer; Sedentary Lifestyle
MeSH Terms: conditions — Colorectal Neoplasms; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the sedentary behavior intervention or the monitoring-only control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary behavior intervention group (Experimental): This group will wear an activity monitor linked to a smartphone app that will send prompts aimed at interrupting prolonged sedentary bouts
  Interventions: Behavioral: Sedentary Behavior; Device: Bluetooth-enabled activity monitor
- Monitoring-only group (Active Comparator): This group will wear a bluetooth-enabled activity monitor but will not be prompted to change behavior
  Interventions: Device: Bluetooth-enabled activity monitor

INTERVENTIONS:
Behavioral: Sedentary Behavior — Messages delivered via smartphone prompting patients to walk after prolonged sedentary behavior bouts are detected via Bluetooth-enabled activity monitor
  Arms: Sedentary behavior intervention group
Device: Bluetooth-enabled activity monitor — Monitoring activity using a Bluetooth-enabled activity monitor

SUMMARY:
The goal of this research is to develop and test a technology-supported intervention to reduce sedentary behavior before and after cancer surgery. Surgical oncology patients are at elevated risk for postoperative complications and readmissions. Sedentary behavior increases markedly after surgery and hospitalization, and reducing sedentary behavior around the time of cancer surgery could reduce risk while also empowering cancer patients to take a more active role in their recovery.

DETAILED DESCRIPTION:
Colorectal or peritoneal cancer patients scheduled for surgical resection (n=60) will be randomized to either the sedentary behavior intervention or monitoring only. The intervention will use a Bluetooth-enabled activity monitor to detect prolonged sedentary bouts, which will prompt a message delivered via smartphone suggesting that patients walk. The intervention will begin at least two weeks prior to scheduled surgery and will continue through the first 30 days at home following hospital discharge. Outcomes will include objective activity and sedentary behavior, patient-reported symptoms and quality of life using standardized instruments, inflammatory biomarkers, and morbidity and hospital readmission 30-days after index discharge.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for curative surgical treatment of metastatic colorectal or peritoneal cancer at UPMC Shadyside
* Ability to stand and walk unassisted prior to surgery
* Identified at least two weeks prior to their scheduled surgery date

Exclusion Criteria:

* Unable to read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Retention | 30 days post-discharge
  Percentage of those enrolled who completed the program
Acceptability | 30-days post-discharge
  Post-intervention interviews will be conducted to assess acceptability of the program
Adherence | 30-days post-discharge
  Percentages of assessments completed and prompts after which steps were detected

SECONDARY OUTCOMES:
Total objective sedentary behavior | Change from baseline to 30 days post-discharge
  A Bluetooth enabled activity monitor worn throughout the study will estimate the total amount of time spent in sedentary behavior per day
Objective physical activity | Change from baseline to 30 days post-discharge
  A Bluetooth enabled activity monitor worn throughout the study will estimate of number of steps/day.
Patient-reported symptoms | Change from baseline to 30 days post-discharge
  Depressive (CES-D) and physical symptom severity (adapted from the MD Anderson Symptom Inventory)
Patient-reported quality of life | Change from baseline to 30 days post-discharge
  Quality of life (FACT)
Inflammatory biomarkers | 2 weeks post-discharge
  Plasma levels of IL-6 and CRP
Morbidity | 30 days post-discharge
  Grade 3-4 surgical complications within 30 days after index hospital discharge will be extracted from medical records
Mean sedentary behavior bout | Change from baseline to 30 days post-discharge
  A Bluetooth enabled activity monitor will be used to estimate mean daily sedentary bout
Maximum sedentary behavior bout | Change from baseline to 30 days post-discharge
  A Bluetooth enabled activity monitor will be used to estimate maximum daily sedentary bout
Readmission | 30 days post-discharge
  Readmissions within 30 days after index hospital discharge will be extracted from medical records

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Low CA, Danko M, Durica KC, Vega J, Li M, Kunta AR, Mulukutla R, Ren Y, Sereika SM, Bartlett DL, Bovbjerg DH, Dey AK, Jakicic JM. A Real-Time Mobile Intervention to Reduce Sedentary Behavior Before and After Cancer Surgery: Pilot Randomized Controlled Trial. JMIR Perioper Med. 2023 Jan 12;6:e41425. doi: 10.2196/41425. PMID 36633893